CLINICAL TRIAL: NCT03996850
Title: SPECT/CT for the Characterization of Renal Masses: Impact on Clinical Decision Making
Brief Title: SPECT/CT for the Characterization of Renal Masses
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-001817; NCI-2019-02711 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Kidney Neoplasm; Renal Mass
MeSH Terms: conditions — Kidney Neoplasms | interventions — X-Rays; Photons; Technetium Tc 99m Sestamibi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health service research (MIBI SPECT/CT, questionnaire): Patients receive technetium Tc-99m sestamibi IV then undergo SPECT/CT.
  Interventions: Procedure: Computed Tomography; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium Tc-99m Sestamibi

INTERVENTIONS:
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Other: Questionnaire Administration — Ancillary studies
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium Tc-99m Sestamibi — Given IV
  Other Names: Cardiolite; Miraluma; Tc 99m Sestamibi; Tc-99m MIBI; Tc99m Sestamibi

SUMMARY:
This trial studies how well technetium Tc-99m sestamibi single-photon emission computed tomography/computed tomography (SPECT/CT) works on clinical decision making in patients with kidney tumors. Diagnostic procedures, such as technetium Tc-99m sestamibi SPECT/CT may be a less invasive way to check for kidney tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of technetium Tc-99m sestamibi (MIBI) SPECT/CT on patient management decisions.

SECONDARY OBJECTIVES:

I. To evaluate the impact of MIBI SPECT/CT on patient management decisions for tumors 1.5-3.0 cm and 3.1-5.0 cm.

II. To assess the impact of MIBI SPECT/CT on decisional conflict score. III. To assess the impact of MIBI SPECT/CT on physician management recommendation.

IV. To evaluate the sensitivity and specificity of MIBI SPECT/CT for the identification of an oncocytic renal mass (oncocytoma, chromophobe, and hybrid oncocytic tumor) with respect to tumor histology identified by renal mass biopsy or surgical resection.

V. To compare the specificity of MIBI SPECT/CT with conventional cross-sectional imaging in predicting an oncocytic renal mass.

VI. To assess the correlation between MIBI SPECT/CT outcomes to final treatment decisions.

EXPLORATORY OBJECTIVES:

I. Evaluate the mitochondria content in tumors that had positive MIBI SPECT/CT findings.

OUTLINE:

Patients receive technetium Tc-99m sestamibi intravenously (IV) then undergo SPECT/CT.

After completion of study, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Performance status Eastern Cooperative Oncology Group (ECOG) < 2.
* Life expectancy (> 1 year).
* New diagnosis of a renal tumor (within past 3 months).
* Measurable, predominantly (> 80%) solid renal neoplasm between 1.5-5.0 cm.
* Lesion concerning for kidney cancer bases on a contrast-enhanced CT or magnetic resonance imaging (MRI).
* No definitive evidence of metastatic disease.
* Does not require urgent surgical treatment.
* Candidate for surgical, ablative, and surveillance approach.
* Willingness to obtain more information to aid decision-making.
* Understanding and willingness to provide consent.

Exclusion Criteria:

* Presence of multiple solid renal tumors.
* A prior needle biopsy of the mass resulting in histologic diagnosis.
* A prior diagnosis of kidney cancer.
* Presence of an active, untreated, non-renal malignancy.
* History of bleeding diathesis or recent bleeding episode.
* Prior surgery or radiation therapy to the kidney.
* Unwillingness to fill out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new diagnosis of a renal tumor (within past 3 months)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient management decision | 6 months
  Assessed with post-test, physician counseling.

SECONDARY OUTCOMES:
Decision making based on tumor size | 6 months
  Could be differentially impacted in two strata, tumors 1.5-3.0 cm and 3.1-5.0 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shuch, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States